CLINICAL TRIAL: NCT05382026
Title: Milk Versus a Pea-based Beverage for Increasing Muscle Mass and Bone Mineral Density During Resistance Training in Adolescent Boys and Girls
Brief Title: Milk Versus a Pea-based Beverage for Bone and Muscle Health in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3228
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1% chocolate milk (Experimental): 250 ml of 1% chocolate milk consumed immediately after resistance training sessions + 250 ml of chocolate milk consumed 1 hour after resistance training sessions
  Interventions: Dietary Supplement: Nutritional supplementation during a 6 month resistance training program
- Pea-based beverage (Active Comparator): 250 ml of pea beverage consumed immediately after resistance training sessions + 250 ml of pea beverage consumed 1 hour after resistance training sessions
  Interventions: Dietary Supplement: Nutritional supplementation during a 6 month resistance training program
- Placebo: Low protein plant-based beverage (Placebo Comparator): 250 ml of placebo beverage consumed immediately after resistance training sessions + 250 ml of placebo beverage consumed 1 hour after resistance training sessions
  Interventions: Dietary Supplement: Nutritional supplementation during a 6 month resistance training program

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation during a 6 month resistance training program — 1% chocolate milk
  Arms: 1% chocolate milk
Dietary Supplement: Nutritional supplementation during a 6 month resistance training program — Pea-based beverage
  Arms: Pea-based beverage
Dietary Supplement: Nutritional supplementation during a 6 month resistance training program — Maltodextrin placebo
  Arms: Placebo: Low protein plant-based beverage

SUMMARY:
Canada's Food Guide places an increased emphasis on plant-based proteins; however, Canadians who consume a plant-based diet may be compromised because of intake of lower-quality protein. Consumption of high-quality protein is important during growth and development, especially in highly active individuals. The study will compare milk (i.e. high quality protein) to a pea-based beverage (i.e. lower quality plant-based protein) in adolescent boys and girls who are engaged in resistance-training programs as part of their athletic training. One-hundred and fourteen adolescent boys and girls (12-17y of age) will be divided into groups that consume milk, a pea-beverage, or a carbohydrate (sugar) beverage after resistance training sessions performed three times per week for six months. It is predicted that the group consuming milk will have greater increases in muscle mass, strength, and bone density, and greater reductions in fat mass compared to the groups consuming a pea-based or carbohydrate beverages.

DETAILED DESCRIPTION:
Milk protein is important especially for very active people and in the context of plant-based diets, which are lower in protein quality. The purpose of the study is to compare the effectiveness of milk supplementation to pea-beverage supplementation during resistance training programs for increasing lean tissue mass in adolescent boys and girls. Secondary and tertiary outcomes include fat mass, bone mineral density, and muscular strength. It is hypothesized that milk supplementation during resistance training will be more effective than plant-based proteins (i.e. pea-beverage) for increasing muscle mass, reducing fat mass, and improving bone mineral outcomes in adolescent boys and girls. One-hundred and fourteen boys and girls (aged 12-17y) who are currently enrolled in resistance training programs (3 times per week for 6 months) as part of their competitive athletic programs will be stratified by sex and maturity status before being randomized to three groups: 1) 1% chocolate milk supplementation; 2) pea-based beverage; 3) carbohydrate beverage (placebo control). Beverages will be consumed during recovery from each resistance training session (i.e. 250 ml immediately after training and 250 ml one hour later to optimize post-exercise protein synthesis) over the six-month intervention. It is anticipated that milk supplementation will be more effective than plant-based protein supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in a resistance-training program 3 times per week
* Female participants must have reached menarche

Exclusion Criteria:

* Have taken any nutritional supplement (e.g., protein, creatine, amino acids) within the past month
* Currently taking anabolic steroids or oral corticosteroids
* Allergies to dairy, almonds, cashews, or peas

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in lean tissue mass (kg) | 6 months
  Lean tissue mass measured by dual energy X-ray absorptiometry

SECONDARY OUTCOMES:
Change in fat mass (kg) | 6 months
  Fat mass measured by dual energy X-ray absorptiometry
Change in lumbar spine bone mineral density (g/cm-squared) | 6 months
  Lumbar spine bone mineral density measured by dual energy X-ray absorptiometry
Change in hip bone mineral density (g/cm-squared) | 6 months
  Hip bone mineral density measured by dual energy X-ray absorptiometry
Change in bench press strength (kg) | 6 months
  Bench press strength predicted from resistance lifted for 6-10 repetitions
Change in squat strength (kg) | 6 months
  Squat strength predicted from resistance lifted for 6-10 repetitions
Change in cross-sectional moment of inertia at the hip (cm to the power of 4) | 6 months
  Cross-sectional moment of inertia measured by dual energy X-ray absorptiometry
Change in section modulus at the hip (cm to the power of 3) | 6 months
  Section modulus measured by dual energy X-ray absorptiometry
Change in cross-sectional area at the hip (cm-squared) | 6 months
  Cross-sectional area measured by dual energy X-ray absorptiometry
Change in cortical thickness at the hip (cm) | 6 months
  Cortical thickness measured by dual energy X-ray absorptiometry
Change in buckling ratio at the hip (no units) | 6 months
  Buckling ratio measured by dual energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No